CLINICAL TRIAL: NCT03614975
Title: Immunologic Response to Influenza Vaccination in Children and Adolescents: A RCT Trial of Influenza Vaccines
Brief Title: Immunologic Response to Influenza Vaccination in Children and Adolescents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Richard Zimmerman MD (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Richard Zimmerman MD, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO18050091; CDCU01IP001035 (Other Grant/Funding Number: Centers for Disease Control and Prevention)
Record Dates: First submitted 2018-06-06; First posted 2018-08-03 (Actual); Results first posted 2019-11-12 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Influenza, Human; Immune Response
Keywords: inactivated; influenza; vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: 1:1 RCT allocation to one of two influenza vaccines: Flucelvax or Fluzone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Flucelvax inactivated influenza vaccine (Active Comparator): Participants receiving inactivated Flucelvax influenza vaccine will receive 0.5 mL given intramuscularly
  Interventions: Biological: Flucelvax inactivated influenza vaccine
- Fluzone inactivated influenza vaccine (Active Comparator): Participants receiving inactivated Fluzone influenza vaccine will receive 0.5 mL given intramuscularly
  Interventions: Biological: Fluzone inactivated influenza vaccine

INTERVENTIONS:
Biological: Flucelvax inactivated influenza vaccine — Participants randomized to this study influenza vaccine arm will receive Flucelvax inactivated influenza vaccine at baseline after the baseline blood draw is complete. (Provided that this vaccine is available clinically in time for the study.)
  Arms: Flucelvax inactivated influenza vaccine
Biological: Fluzone inactivated influenza vaccine — Participants randomized to this study influenza vaccine arm will receive Fluzone inactivated influenza vaccine at baseline after the baseline blood draw is complete. (Provided that this vaccine is available clinically in time for the study.)
  Arms: Fluzone inactivated influenza vaccine

SUMMARY:
The purpose of this study is to evaluate immunologic response to different types of influenza vaccine among children/adolescents/young adults 4-20 years of age. This is a randomized controlled trial (RCT), that will assess immune response in 120 participants (60 per vaccine arm) pre- and post-vaccination to Flucelvax (egg-free inactivated flu shot) and Fluzone (egg-based inactivated flu shot).

DETAILED DESCRIPTION:
This is a non-blinded, randomized controlled trial analyzing influenza vaccine immunogenicity response in children/adolescents/young adults aged 4-20 years given one of two FDA approved and licensed influenza vaccines: Flucelvax (egg-free inactivated flu shot) and Fluzone (egg-based inactivated flu shot). This study will enroll 120 healthy participants, 60 per vaccine arm. Participants will be randomized using a 1:1 allocation to receive either Flucelvax or Fluzone. Blood work will be conducted on all participants at baseline prior to vaccine receipt and post-vaccination at Day 7 (range 6-9 days) and Day 21 (range 21-35 days). The primary objective of the study is to determine pre and post serologic,responses to each vaccine type.

ELIGIBILITY:
Inclusion Criteria:

* aged 4-20 years;
* has prior vaccination history available (which can be determined based either on medical record review or through state registry review;
* plans to receive the current seasonal influenza vaccination at one of the recruiting sites

Exclusion Criteria:

* unable or unwilling to completed required study activities, including informed consent, randomization to vaccine, and bloodwork;
* has already received influenza vaccine for the current season;
* has a known immunocompromising condition or is on an immunosuppressing medication (e.g., high dose steroids >10 days);
* is known to be pregnant;
* has a history of severe allergy to eggs or to influenza vaccine or any of its components

Ages: 4 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 166 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2018-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard K Zimmerman, MD, MPH, MA, Principal Investigator — University of Pittsburgh, School of Medicine, Dept. Family Medicine
Locations (2):
- United States (2):
  - General Academic Pediatrics, Pittsburgh, Pennsylvania
  - University of Pittsburgh Department of Family Medicine, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the primary article, after deidentification, will be placed at the site mentioned below.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months after article publication.
Access Criteria: Researchers who provide a methodologically sound proposal and have appropriate data security and privacy plans in place
URL: https://github.com/pittvax

REFERENCES:
- [Derived] Moehling KK, Zimmerman RK, Nowalk MP, Jeng Lin C, Martin JM, Alcorn JF, Susick M, Burroughs A, Holiday C, Flannery B, Levine MZ. A randomized controlled trial of antibody response to 2018-19 cell-based vs. egg-based quadrivalent inactivated influenza vaccine in children. Vaccine. 2020 Jul 14;38(33):5171-5177. doi: 10.1016/j.vaccine.2020.06.023. Epub 2020 Jun 21. PMID 32580919

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Flucelvax Inactivated Influenza Vaccine | Fluzone Inactivated Influenza Vaccine
Started | 85 | 81
Completed | 75 | 73
Not Completed | 10 | 8
Not completed — Physician Decision | 7 | 5
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Specimens not in lab batch shipment | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flucelvax Inactivated Influenza Vaccine | Fluzone Inactivated Influenza Vaccine | Total
Number analyzed (Participants) | 85 | 81 | 166
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Only subjects who completed the study to day 21 were included in this analysis
  years
    number analyzed (Participants) | 75 | 73 | 148
    (all) | 14.03 [10.77 to 15.88] | 14.21 [11.46 to 16.60] | 14.07 [10.91 to 16.21]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only participants who completed the study through day 21 were included in this analysis
  Participants
    number analyzed (Participants) | 75 | 73 | 148
    Female | 39 | 40 | 79
    Male | 36 | 33 | 69
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only data on participants who completed day 21 of the study are reported.
  Participants
    number analyzed (Participants) | 75 | 73 | 148
    American Indian or Alaska Native | 0 | 1 | 1
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Black or African American | 53 | 50 | 103
    White | 14 | 14 | 28
    More than one race | 7 | 7 | 14
    Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 85 | 81 | 166

OUTCOME MEASURES:

1. Primary Outcome: Determining Seroconversion Response - Change in HI Titers From Pre- to Post Vaccination
Description: Hemagglutination inhibition (HI) assay will be conducted to assess immunologic outcome. Seroconversion is defined as a 4-fold or higher rise in HI titer post-vaccination given a pre-vaccination HI titer of >= 10.
Time Frame: Pre-vaccination (at Day 0 timepoint) and post-vaccination (at Day 21 timepoint)
Population: Participants who completed study through day 21
Measure: Count of Participants; unit: Participants
Arm/Group | Flucelvax Inactivated Influenza Vaccine | Fluzone Inactivated Influenza Vaccine
Number analyzed (Participants) | 75 | 73
Participants
  Vaccine Strain: A/H1N1 | 20 | 14
  Vaccine Strain: A/H3N2 | 9 | 11
  Vaccine Strain: B/Colorado | 22 | 24
  Vaccine Strain: B/Phuket | 14 | 9
Statistical Analysis 1: Comparison: Flucelvax Inactivated Influenza Vaccine vs Fluzone Inactivated Influenza Vaccine; Test type: Other; p = 0.28, Chi-squared — A/H1N1
Statistical Analysis 2: Comparison: Flucelvax Inactivated Influenza Vaccine vs Fluzone Inactivated Influenza Vaccine; Test type: Other; p = 0.64, Chi-squared — A/H3N2
Statistical Analysis 3: Comparison: Flucelvax Inactivated Influenza Vaccine vs Fluzone Inactivated Influenza Vaccine; Test type: Other; p = 0.64, Chi-squared — B/Colorado
Statistical Analysis 4: Comparison: Flucelvax Inactivated Influenza Vaccine vs Fluzone Inactivated Influenza Vaccine; Test type: Other; p = 0.23, Chi-squared — B/Phuket

2. Secondary Outcome: Determining Seroprotection Level at Each Time Point
Description: Hemagglutination inhibition assay will be conducted to assess immunologic outcome. Seroprotection is defined as a HI titer >= 1:110 at either time point.
Time Frame: Pre-vaccination (at Day 0 timepoint) and post-vaccination (at Day 21 timepoint)
Population: Data was analyzed on participants who completed day 21 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Flucelvax Inactivated Influenza Vaccine | Fluzone Inactivated Influenza Vaccine
Number analyzed (Participants) | 75 | 73
Participants
  Vaccine Strain: A/H1N1 : Day 0 | 45 | 39
  Vaccine Strain: A/H1N1 : Day 21 | 66 | 58
  Vaccine Strain: A/H3N2 : Day 0 | 51 | 45
  Vaccine Strain: A/H3N2 : Day 21 | 62 | 60
  Vaccine Strain: B/Colorado : Day 0 | 37 | 35
  Vaccine Strain: B/Colorado : Day 21 | 56 | 56
  Vaccine Strain: B/Phuket : Day 0 | 48 | 41
  Vaccine Strain: B/Phuket : Day 21 | 61 | 53
Statistical Analysis 1: Comparison: Flucelvax Inactivated Influenza Vaccine vs Fluzone Inactivated Influenza Vaccine; Test type: Other; p = 0.42, Chi-squared — Vaccine Strain: A/H1N1:Day 0
Statistical Analysis 2: Comparison: Flucelvax Inactivated Influenza Vaccine vs Fluzone Inactivated Influenza Vaccine; Test type: Other; p = 0.16, Chi-squared — Vaccine Strain: A/H1N1: Day 21
Statistical Analysis 3: Comparison: Flucelvax Inactivated Influenza Vaccine vs Fluzone Inactivated Influenza Vaccine; Test type: Other; p = 0.42, Chi-squared — Vaccine Strain: A/H3N2: Day 0
Statistical Analysis 4: Comparison: Flucelvax Inactivated Influenza Vaccine vs Fluzone Inactivated Influenza Vaccine; Test type: Other; p = 0.94, Chi-squared — Vaccine Strain: A/H3N2: Day 21
Statistical Analysis 5: Comparison: Flucelvax Inactivated Influenza Vaccine vs Fluzone Inactivated Influenza Vaccine; Test type: Other; p = 0.87, Chi-squared — Vaccine Strain: B/Colorado :Day 0
Statistical Analysis 6: Comparison: Flucelvax Inactivated Influenza Vaccine vs Fluzone Inactivated Influenza Vaccine; Test type: Other; p = 0.77, Chi-squared — Vaccine Strain: B/Colorado : Day 21
Statistical Analysis 7: Comparison: Flucelvax Inactivated Influenza Vaccine vs Fluzone Inactivated Influenza Vaccine; Test type: Other; p = 0.33, Chi-squared — Vaccine Strain: B/Phuket: Day 0
Statistical Analysis 8: Comparison: Flucelvax Inactivated Influenza Vaccine vs Fluzone Inactivated Influenza Vaccine; Test type: Other; p = 0.21, Chi-squared — Vaccine Strain: B/Phuket: Day 21

3. Secondary Outcome: Determining Geometric Mean Titers (GMTs) at Each Time Point
Description: Hemagglutination inhibition assay will be conducted to assess immunologic outcome. GMTs is defined as the anti-log of the mean of the log2 HI titers
Time Frame: Pre-vaccination (at Day 0 timepoint) and post-vaccination (at Day 21 timepoint)
Measure: Geometric Mean (95% Confidence Interval); unit: Dilution
Arm/Group | Flucelvax Inactivated Influenza Vaccine | Fluzone Inactivated Influenza Vaccine
Number analyzed (Participants) | 75 | 73
Dilution
  Vaccine Strain: A/H1N1 : Day 0 | 6.63 [6.29 to 7.01] | 6.42 [6.05 to 6.82]
  Vaccine Strain: A/H1N1 : Day 21 | 8.08 [7.82 to 8.36] | 7.76 [7.46 to 8.08]
  Vaccine Strain: A/H3N2 : Day 0 | 7.42 [7.16 to 7.69] | 6.94 [6.58 to 7.32]
  Vaccine Strain: A/H3N2 : Day 21 | 7.90 [7.63 to 8.18] | 7.96 [7.70 to 8.22]
  Vaccine Strain: B/Colorado : Day 0 | 6.55 [6.19 to 6.93] | 6.42 [6.03 to 6.83]
  Vaccine Strain: B/Colorado : Day 21 | 7.56 [7.21 to 7.92] | 7.71 [7.39 to 8.05]
  Vaccine Strain: B/Phuket : Day 0 | 6.78 [6.43 to 7.15] | 6.52 [6.16 to 6.91]
  Vaccine Strain: B/Phuket : Day 21 | 7.34 [7.01 to 7.69] | 7.46 [7.11 to 7.80]
Statistical Analysis 1: Comparison: Flucelvax Inactivated Influenza Vaccine vs Fluzone Inactivated Influenza Vaccine; Test type: Other; p = 0.49, Kruskal-Wallis — Vaccine Strain: A/H1N1: Day 0
Statistical Analysis 2: Comparison: Flucelvax Inactivated Influenza Vaccine vs Fluzone Inactivated Influenza Vaccine; Test type: Other; p = 0.23, Kruskal-Wallis — Vaccine Strain: A/H1N1: Day 21
Statistical Analysis 3: Comparison: Flucelvax Inactivated Influenza Vaccine vs Fluzone Inactivated Influenza Vaccine; Test type: Other; p = 0.10, Kruskal-Wallis — Vaccine Strain: A/H3N2: Day 0
Statistical Analysis 4: Comparison: Flucelvax Inactivated Influenza Vaccine vs Fluzone Inactivated Influenza Vaccine; Test type: Other; p = 0.86, Kruskal-Wallis — Vaccine Strain: A/H3N2: Day 21
Statistical Analysis 5: Comparison: Flucelvax Inactivated Influenza Vaccine vs Fluzone Inactivated Influenza Vaccine; Test type: Other; p = 0.73, Kruskal-Wallis — Vaccine Strain: B/Colorado: Day 0
Statistical Analysis 6: Comparison: Flucelvax Inactivated Influenza Vaccine vs Fluzone Inactivated Influenza Vaccine; Test type: Other; p = 0.67, Kruskal-Wallis — Vaccine Strain: B/Colorado: Day 21
Statistical Analysis 7: Comparison: Flucelvax Inactivated Influenza Vaccine vs Fluzone Inactivated Influenza Vaccine; Test type: Other; p = 0.36, Kruskal-Wallis — Vaccine Strain: B/Phuket: Day 0
Statistical Analysis 8: Comparison: Flucelvax Inactivated Influenza Vaccine vs Fluzone Inactivated Influenza Vaccine; Test type: Other; p = 0.65, Kruskal-Wallis — Vaccine Strain: B/Phuket: Day 21

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Flucelvax Inactivated Influenza Vaccine | Fluzone Inactivated Influenza Vaccine
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/81
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/81
Other Adverse Events (participants affected / at risk) | 0/85 | 0/81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/75/NCT03614975/Prot_SAP_000.pdf